CLINICAL TRIAL: NCT04892056
Title: Evaluation of the Rate of Anterior Segment Retraction Using Friction Versus Frictionless Mechanics: A Randomized Clinical Trial
Brief Title: Evaluation of the Rate of Anterior Segment Retraction Using Two Types of Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Monica Guirguis Youssif Tawfik, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FUE.REC 9/10-2018
Record Dates: First submitted 2021-04-27; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Bimaxillary Protrusion
Keywords: T loops; Friction; Frictionless; power chains; digital models; anterior segment retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the principal investigator was not possible due to the nature of the interventions. However, the outcome assessor was blinded to the interventions and all digital models were unidentified during outcome assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Segment Retraction using Friction mechanics by elastomeric power chains (Experimental): Elastomeric power chains extending from 8mm crimpable hooks, distal to the lateral incisors, on 0.017"x0.025" Stainless Steel WIres, to the mini-screws. The power chains delivered 160g of force per side.
  Interventions: Other: Friction Mechanics
- Anterior Segment Retraction using Frictionless mechanics by T-loops (Experimental): T shaped closing loops were fabricated on 0.017"x0.025" Titanium- Molybdenum wires (TMA) were used to deliver 160g of force per side by 4mm distal activations.
  Interventions: Other: Frictionless Mechanics

INTERVENTIONS:
Other: Friction Mechanics — anterior segment retraction using elastomeric power chains
  Other Names: sliding mechanics
  Arms: Anterior Segment Retraction using Friction mechanics by elastomeric power chains
Other: Frictionless Mechanics — anterior segment retraction using closing loops
  Other Names: segmented mechanics
  Arms: Anterior Segment Retraction using Frictionless mechanics by T-loops

SUMMARY:
The rate of anterior segment retraction in bi-maxillary protrusion cases was evaluated comparing the friction and friction-less mechanics. since, there has been a lack of clear cut guidelines for clinicians for the optimum method for retraction, this randomized clinical trial was done.

DETAILED DESCRIPTION:
Thirty bi-maxillary protrusion female patients were randomly allocated into either intervention groups. In the Friction group, retraction was accomplished using elastomeric power chains extending from crimpable hooks distal to the lateral incisors, on 0.017x0.025-inch Stainless Steel wires, to the mini-screws . While in the friction-less group with retraction done using T- loop springs made of 0.017x0.025-inch titanium molybdenum wires. Retraction force was set to 160g per side in both intervention groups. Activation was done every four weeks. Rate of anterior segment retraction was evaluated via digital models.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects.
* Age 13-25 y of age.
* Skeletal Angle Class I malocclusion with Bimaxillary dentoalveolar protrusion in need of four 1st premolar extractions with maximum anchorage.
* Fully erupted permanent dentition without crowding.
* Good oral and general health.

Exclusion Criteria:

* Systemic Diseases or syndromes or on anti-inflammatory medication.
* Extracted or missing permanent teeth.
* History of previous Orthodontic Treatment.
* Parafunctional Habits.
* Badly decayed teeth.

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of Anterior Segment Retraction | The start of anterior segment retraction up to complete space closure, an average of 6 months.
  The rate of anterior segment retraction per month was measured on monthly digital models.

SECONDARY OUTCOMES:
Anchorage Loss | The start of anterior segment retraction up to complete space closure, an average of 6 months.
  Mesial movement of the first primary molar was evaluated on the digital models
Pain experienced after each activation of the two mechanics | The start of anterior segment retraction up to complete space closure, an average of 6 months.
  Patients were asked to complete Visual Analogue Scales of the degree of pain after every intervention. The scale values between 0 to 10, with 0 being no pain experienced by the patient and 10 being the highest level of pain experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, Chairman, Study Chair — Future Univeristy in Egypt
Locations (1):
- Future Univeristy in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After Publication

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT04892056/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT04892056/ICF_001.pdf